CLINICAL TRIAL: NCT06120946
Title: The Influence of Cerebral Protection on Neurocognitive Outcomes Following Transcatheter Aortic Valve Implantation (TAVI)
Brief Title: Neurocognitive Assessment in TAVI
Acronym: NEAT TAVI
Status: Completed | Type: Observational
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Collaborators: University of Melbourne (Other); Terumo Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: NEAT TAVI
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control arm: Patients randomised in the BHF PROTECT study to TAVI without Sentinel cerebral embolic protection
- Intervention arm: Patients randomised in the BHF PROTECT study to TAVI with Sentinel cerebral embolic protection

SUMMARY:
Severe aortic stenosis is a common heart condition affecting elderly patients. Degeneration of the aortic valve (oneway valve between the heart and the aorta) causes high resistence to blood flow, resulting in strain on the heart and the potential for heart failure and death. Treatment of aortic stenosis has traditionally been with open heart surgery. A new procedure called transcatheter aortic valve implantation (TAVI) allows new aortic valves to be implanted through the femoral arteries, resulting in equivalent outcomes to open surgery with a more rapid recovery. Some complications remain present however, including the risk of debris released during the valve implantation being carried by the blood stream into the brain. This may lead to strokes and a loss of mental capacity. Devices that filter the blood stream and capture this debris have now been developed but are of uncertain benefit. We plan to investigate the brain function of patients who have been randomly assigned to the TAVI procedure with and without the use of filters to see if there are any cognitive benefits to the use of this technology.

Patients who are enrolled in the BHF PROTECT-TAVI trial will be invited to partcipate in this trial. They will have already been randomly assigned to TAVI with or without cerebral filter use. We will perform a series of bedside clinical tests (lasting ~40 minutes) involving questionnaires, pen & paper and computer-based tasks. These will be performed both pre- and post-TAVI. There is no change to routine patient care. Data will be analysed with the assistance of trained neuropsychologists and will provide a valuable insight into the performance and role of the cerebral filter for TAVI patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Randomised in the BHF PROTECT-TAVI trial (assessing stroke outcomes in TAVI with and without filter use).
* Willing to provide informed consent for participation in this trial.

Exclusion Criteria:

* Participant has been excluded from use of the filter device due to anatomical or clinical contra-indications.
* Inadequate English skills.
* Inability to complete assessment tasks due to visual or auditory impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from those undergoing Transcatheter Aortic Valve Implantation at the Royal Sussex County Hospital, Brighton, United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Neurocognitive change | <3 days post-TAVI
  Neurocognitive change by individual scores for each task performed

SECONDARY OUTCOMES:
Neurocognitive change | 12-months post-TAVI
  Neurocognitive change by individual scores for each task performed

OTHER OUTCOMES:
Subgroup interactions | <3 days post-TAVI
  Age, baseline cognitive score, prior CVA, type of TAVI device, procedural pre- and post-dilation

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Sussex County Hospital, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Pending based on BHF PROTECT study